CLINICAL TRIAL: NCT02545751
Title: A Phase II Study of Stereotactic Body Radiation Therapy and ZADAXIN's® (Thymalfasin) Induced Tumor Effects in Patients With Heavily Pretreated, Metastatic Esophageal Cancer
Brief Title: SBRT Combined With Thymalfasin for Metastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shixiu Wu, MD, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hangzhou CH
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Esophageal Cancer; Metastatic Esophageal Cancer; Stereotactic Body Radiation Therapy; Thymalfasin
Keywords: Esophageal cancer; Metastatic esophageal cancer; Radiotherapy; Thymalfasin; ZADAXIN's®; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiosurgery; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT and Thymalfasin arm (Experimental): SBRT is given during combined therapy to one of the lesions, 25Gy in 5 fractions over one week, conformally to maximally spare normal tissue or organ. Thymalfasin treatment is given twice a week with an interval of 3-4 days until tumor progression of other metastatic lesions. Tumor response is evaluated by assessing clinical and CT/MRI response for all the other measurable metastatic sites.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Drug: Thymalfasin

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT is given during combined therapy to one of the metastatic lesions, 25Gy in 5 fractions (5Gy per fraction) over one week, conformally to maximally spare normal tissue or organ.
  Other Names: SBRT
Drug: Thymalfasin — Thymalfasin treatment is given twice a week with an interval of 3-4 days until progression of other metastatic lesions. Tumor response is evaluated by assessing clinical and CT/MRI response for all the other measurable metastatic sites.
  Other Names: ZADAXIN's®

SUMMARY:
Patients with esophageal cancer that had metastatic lesions after been treated with definitive surgery or chemoradiotherapy are being asked to participate in this study.

1. To observe immunity-mediated tumor response after Stereotactic Body Radiation Therapy(SBRT) of a metastatic site in metastatic esophageal cancer patients.
2. To induce the efficacy (effectiveness) of a new combination of therapy, SBRT and thymalfasin for heavily pretreated, metastatic esophageal cancer patients; This study will help find out what effects (good or bad) the combination of radiotherapy and thymalfasin has on metastatic esophageal cancer.

DETAILED DESCRIPTION:
1. To observe immunity-mediated tumor response after Stereotactic Body Radiation Therapy(SBRT) of a metastatic site in metastatic esophageal cancer patients.
2. To induce the efficacy (effectiveness) of a new combination of therapy, SBRT and thymalfasin for heavily pretreated, metastatic esophageal cancer patients; Eligible are patients with metastatic esphageal cancer who have achieved stable disease or have disease progression after systemic therapy (surgery or definitive chemoradiotherapy) and have at least two measurable sites of metastatic lesions. Extent of metastatic disease is recorded both at CT and PET/CT scanning. Radiation is given during combined therapy to one of the lesions, 25Gy in 5 fractions over one week interval with SBRT, conformally to maximally spare normal tissue or organ. Thymalfasin treatment is given twice a week with an interval of 3-4 days each week for a total of 8 weeks. Tumor response is evaluated by assessing clinical and CT/MRI response for all of the measurable metastatic sites. A Phase II clinical trial based on an optimum two-stage Phase II Simon design is used to conduct this pilot study. Ten patients will be treated in Stage one; if there are no tumor responses, the trial will be terminated. If there are one or more tumor responses in Stage One, the trial will proceed to enroll an additional 19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed esophageal cancer which is persistent and metastatic or recurrent and metastatic;
2. Patients must have at least 2 distinct measurable metastatic sites at least 1 cm of larger in their largest diameter;
3. Age ≥18 years;
4. Metastatic disease measurable on a CT/MRI scan. The primary tumor is not considered measurable disease. Metastatic lesions within a prior radiation field are acceptable as long as disease has progressed in the radiation field by RECIST criteria. The same imaging modality performed at baseline (CT or MRI) will be repeated at subsequent imaging.
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Patients have adequate baseline organ and marrow function as defined by an absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Signed consent forms voluntarily;

Exclusion Criteria:

1. Patients undergoing therapy with other investigational agents.
2. Women who are pregnant or breastfeeding;
3. Patients with known brain metastases can be included in this clinical trial but brain lesions are not eligible as target or non target lesion;
4. Anticipated patient survival under 3 months;
5. Active severe infection or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus;
6. Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, myocardial infarction, stroke or congestive heart failure within the last 6 months;
7. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
8. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
9. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with tumor responses after the initiation of treatment. | month 1- month 6

SECONDARY OUTCOMES:
The number of participants with adverse events from the date of enrollment until 2 years from the opening of the study. | year 0- year 2
The proportion of patients alive with tumor responses from the date of enrollment until date of death from any cause, assessed up to 2 years from the opening of the study. | year 0- year 2

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, MD, Study Chair — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China